CLINICAL TRIAL: NCT02489773
Title: Lucica ® Glycated Albumin-L Clinical Program - Pivotal Study
Status: Completed | Type: Observational
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP002
Record Dates: First submitted 2015-06-15; First posted 2015-07-03 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Diabetes
Keywords: Lucica; glycated albumin; GA; fructosamine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: HbA1c values ranged from 7.5% to 12% (or higher)
- Group 2: HbA1c values <7.5%

SUMMARY:
To confirm that Lucica ® Glycated Albumin-L is useful for the intermediate term (preceding 2-3 weeks) monitoring of glycemic control in patients with diabetes.

DETAILED DESCRIPTION:
In order to confirm that Lucica ® Glycated Albumin-L is useful for the intermediate term (preceding 2-3 weeks) monitoring of glycemic control in patients with diabetes, subjects with Type 1 or Type 2 diabetes will be enrolled whose HbA1c values range from 7.5% to 12% (or higher) in Group 1 and <7.5% in Group 2 at Visit 1, and the comparison of glycated albumin (GA) and other glycemic control indices will be performed during 6 months in 8 clinical sites in US. Group 1 will consist of 90 evaluable subjects who have a change in diabetes management to improve glycemic control; this therapy can include oral agents, insulin, or noninsulin injectable anti-diabetic medications. Group 2 will consist of 40 evaluable subjects already on a stable diabetic management program, who have had no change in treatment in the last 3 months and for whom there is no plan to make a change during the study period.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study if they meet all the following criteria:

1. Male and female subjects 18 years of age and older
2. Subjects with Type 1 or Type 2 diabetes (enrolled in an approximate ratio of 1:1, respectively)
3. Subjects with an HbA1c value within the range of 7.5% to 12% (or higher) for Group 1 and <7.5% for Group 2

   Note: The study investigator or primary physician must be planning to institute, or must be in the process of instituting, therapy to improve glycemic control for subjects in Group 1; this therapy can include oral agents, insulin, or non-insulin injectable anti-diabetic medications.
4. Willingness to complete the protocol requirements, including the use of self-monitoring of blood glucose (SMBG) and attendance at all scheduled study visits; if selected for continious glucose monitoring (CGM) , a willingness to follow the additional requirements and to use only the CGM device model provided for the study
5. Satisfactory completion of home SMBG measurements during the screening period of the study prior to enrollment at Visit 2

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Any clinically significant disease, as determined by the investigator, that would interfere with study evaluations including but not limited to the following current or historical conditions/procedures (self-reported by the subject):

   1. End-stage renal disease
   2. Chronic kidney disease of Stage 3 or greater
   3. Liver cirrhosis
   4. Uncontrolled or untreated thyroid disease
   5. Any other acute or chronic conditions that, in the opinion of the investigator, may significantly influence albumin or glucose metabolism (Note: routine iron deficiencies and abnormal hemoglobin variants are not exclusions)
2. History within the last 6 months of a blood transfusion
3. Any other condition or factor that, in the opinion of the investigator, would complicate or compromise the study or the well-being of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The observational study will include a cross-section of subjects from the intended use population who are being monitored for glycemic control. Equal numbers of subjects with Type 1 or Type 2 diabetes will be enrolled whose HbA1c values range from 7.5% to 12% (or higher) in Group 1 and <7.5% in Group 2 at Visit 1. Group 1 will consist of 90 evaluable subjects who have a change in diabetes management to improve glycemic control; this therapy can include oral agents, insulin, or noninsulin injectable anti-diabetic medications. Group 2 will consist of 40 evaluable subjects already on a stable diabetic management program, who have had no change in treatment in the last 3 months and for whom there is no plan to make a change during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hideji Hiraoka, M.S., Study Director — Diagnostics Department, Asahi Kasei Pharma
Locations (8):
- United States (8):
  - National Research Institute - Huntington Park, Los Angeles, California
  - National Research Institute-Westlake, Los Angeles, California
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Texas Diabetes & Endocrinology, P.A. -Austin, Austin, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Capital Clinical Research Center, Olympia, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Desouza CV, Rosenstock J, Kohzuma T, Fonseca VA. Glycated Albumin Correlates With Time-in-Range Better Than HbA1c or Fructosamine. J Clin Endocrinol Metab. 2023 Oct 18;108(11):e1193-e1198. doi: 10.1210/clinem/dgad298. PMID 37259605
- [Derived] Desouza CV, Holcomb RG, Rosenstock J, Frias JP, Hsia SH, Klein EJ, Zhou R, Kohzuma T, Fonseca VA. Results of a Study Comparing Glycated Albumin to Other Glycemic Indices. J Clin Endocrinol Metab. 2020 Mar 1;105(3):677-87. doi: 10.1210/clinem/dgz087. PMID 31650161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, multicenter, comparative, pivotal study of assay performance in the clinical setting. The target population for this study included up to 150 patients placed into 2 groups, each containing approximately equal numbers of patients with Type 1 or Type 2 diabetes.
Pre-assignment Details: A total of 165 patients were screened for the study, 150 patients were enrolled.
Groups:
- HbA1c Values Ranged From ≥7.5% to 12% (or Higher): Group 1 consisted of at least 90 patients whose HbA1c values ranged from ≥7.5% to 12% (or higher) at screening (Visit 1) and who were prescribed a change in diabetes management to improve glycemic control (therapy could have included oral agents, insulin, or noninsulin injectable anti-diabetic medications).
- HbA1c Values <7.5%: Group 2 consisted of at least 40 patients with HbA1c values <7.5% at Visit 1 who were already on a stable diabetic management program, had no change in treatment in the 3 months prior to screening, and for whom no change was planned during the study period.
Period: Overall Study
Arm/Group | HbA1c Values Ranged From ≥7.5% to 12% (or Higher) | HbA1c Values <7.5%
Started | 98 | 52
Completed | 91 | 50
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Leave the country or the state | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 consisted of at least 90 patients whose HbA1c values ranged from ≥7.5% to 12% (or higher) at screening (Visit 1) and who were prescribed a change in diabetes management to improve glycemic control (therapy could have included oral agents, insulin, or noninsulin injectable anti-diabetic medications).
- Group 2: Group 2 consisted of at least 40 patients with HbA1c values <7.5% at Visit 1 who were already on a stable diabetic management program, had no change in treatment in the 3 months prior to screening, and for whom no change was planned during the study period.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 98 | 52 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (15.61) | 50.3 (15.81) | 50.5 (15.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 27 | 80
  Male | 45 | 25 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 7 | 29
  Not Hispanic or Latino | 76 | 45 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 4 | 17
  White | 80 | 46 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 98 | 52 | 150

OUTCOME MEASURES:

1. Primary Outcome: Compare the Pearson Correlation of Glycated Albumin (GA) and Fructosamine Within All Subjects With the Performance Goal of 0.8
Time Frame: From baseline to 6 months
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | HbA1c Values Ranged From ≥7.5% to 12% (or Higher) | HbA1c Values <7.5%
Number analyzed (Participants) | 98 | 52
Pearson correlation coefficient | 0.7056 | 0.5271
Statistical Analysis 1: Comparison: HbA1c Values Ranged From ≥7.5% to 12% (or Higher) vs HbA1c Values <7.5%; Test type: Other — Calculate the pearson correlation within whole subjects (across Group 1 and Group 2); pearson correlation coefficient = 0.6342
Statistical Analysis 2: Comparison: HbA1c Values Ranged From ≥7.5% to 12% (or Higher) vs HbA1c Values <7.5%; Test type: Other — Diffenrence between Pearson correlations within whole subjects (accross Group 1 and Group 2) and PG, 0.8; p > 0.9999, t-test, 2 sided; Difference with PG 0.8 = -0.1658, 95% CI 2-sided [-0.2204 to -0.1113]

2. Secondary Outcome: Spearman Correlation Analysis of Changes in GA, HbA1c, and 7-day Interval Mean Blood Glucaose (MBG) in the First 3 Months in Group 1
Description: Comparing the Spearman correlation of changes in GA and MBG to the Spearman correlation of changes in HbA1c and MBG, from baseline to any matching post-baseline visit in the first 3 months in Group 1.
Time Frame: From baseline to the first 3 months after enrollment in Group 1
Population: It is pre-specified to collect and report data for only participants who had a change in treatment (Group 1).
Measure: Number; unit: spearman correlation coefficient
Arm/Group | HbA1c Values Ranged From ≥7.5% to 12% (or Higher)
Number analyzed (Participants) | 98
spearman correlation coefficient
  Correlation coefficent between GA and MBG | 0.481
  Correlation coefficent between HbA1c and MBG | 0.233
Statistical Analysis 1: Comparison: HbA1c Values Ranged From ≥7.5% to 12% (or Higher); Test type: Other — The difference in Spearman correlation coefficient between GA and MBG vs HbA1c and MBG in the first 3-month period in Group 1; p < 0.0001, t-test, 2 sided; Difference in correlation coefficients = 0.249, 95% CI 2-sided [0.130 to 0.364]

3. Secondary Outcome: Kendall Correlation Analysis of Changes in GA, HbA1c, and 7-day Interval MBG in the First 3 Months in Group 1
Description: Comparing the Kendall correlation of changes in GA and MBG to the Kendall correlation of changes in HbA1c and MBG, from baseline to any matching post-baseline visit in the first 3 months in Group 1.
Time Frame: From baseline to the first 3 months after enrollment in Group 1
Population: It is pre-specified to collect and report data for only participants who had a change in treatment (Group 1)
Measure: Number; unit: kendall correaltion coefficient
Arm/Group | HbA1c Values Ranged From ≥7.5% to 12% (or Higher)
Number analyzed (Participants) | 98
kendall correaltion coefficient
  Correlation coefficient betwenn GA and MBG | 0.341
  Correlation coefficient betwenn HbA1c and MBG | 0.160
Statistical Analysis 1: Comparison: HbA1c Values Ranged From ≥7.5% to 12% (or Higher); Test type: Other — The difference in Kendall correlation coefficient between GA and MBG vs HbA1c and MBG in the first 3-month period in Group 1; p < 0.0001, t-test, 2 sided; Difference in correlation coefficient = 0.181, 95% CI 2-sided [0.096 to 0.265]

ADVERSE EVENTS:
Time Frame: Adverse events collected from enrolment (6 months)
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/52
Serious Adverse Events (participants affected / at risk) | 5/98 | 3/52
Other Adverse Events (participants affected / at risk) | 53/98 | 28/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=98) | Group 2 (N=52)
A loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Skin ulcea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=98) | Group 2 (N=52)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3)
Gastroenteritis (Infections and infestations) | 7 (7) | 0 (0)
Sinusitis (Infections and infestations) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Paraesthesia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chloelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Planer fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Attention deficit/ Hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After (a) the date multicenter publication is made, (b) Sponsor notifies Institution that there will be no multicenter publication, or (c) 12 months after the date the Study has been closed at all participating sites, whichever date comes first, Institution may itself publish the results of its data from the Study.